CLINICAL TRIAL: NCT05661396
Title: Development of a Therapeutic Serious Game in the Rehabilitation of Stroke Patient
Brief Title: Therapeutic Serious Game and Rehabilitation of Stroke Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopitaux de Saint-Maurice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSU-SG 5
Record Dates: First submitted 2022-11-21; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Stroke; Unilateral Spatial Neglect
Keywords: serious game; stroke; unilateral spatial neglect; rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Behavioral: Serious game rehabilitation
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Serious game rehabilitation — Three patients received therapeutic serious game rehabilitation in addition to conventional rehabilitation. The serious game was proposed to be played three times per week for four weeks, for a total of 12 sessions, with 15 min per session (= 45 minutes per week).
  Arms: Experimental group

SUMMARY:
The growing field of new technologies offers new perspectives for neurorehabilitation. Serious games are a promising solution in the rehabilitation of cognitive impairments, and they may be useful in the rehabilitation of unilateral spatial neglect. The investigators developed a rehabilitation program for visual exploration training with a serious game and investigated its efficiency.

Six patients with unilateral spatial neglect after a right hemispheric stroke were recruited. Three patients assigned to the experimental group received both serious game training and conventional rehabilitation, and three assigned to the control group received only conventional rehabilitation. The investigators compared the two groups after rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral spatial neglect syndrome
* Right cerebral lesion

Exclusion Criteria:

* Epilepsia
* General mental deterioration
* Psychiatric disorder
* No prior history of neurological disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2017-06-03 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Bells test | up to 4 weeks
  35 bells are spatially distributed among distractors on sheet of paper (15 on the left side, 5 on the center and 15 on the right side). Subjects have to cancel as many bells as possible. The number of omissions on the left and on the right side is recorded.

SECONDARY OUTCOMES:
Bisection of lines | up to 4 weeks
  2 lines of 200 millimeters are presented on a sheet of paper. Subjects have to mark the middle of the lines. The deviation from the objective middle is measured in millimeter.
Ogden scene copying | up to 4 weeks
  Copying of the 'Ogden scene' required participants to copy a scene that consisted of 2 trees, a fence and a house (shown from left to right side of the page). Each stroke in the scene to be copied was counted as a point; each omitted stroke was scored as one error, and each distorted or misplaced stroke was scored as one-half of an error (/4).
Reading task | up to 4 weeks
  A text of 116 words is presented with 61 words on the left side and 55 on the right side. Subjects have to read this text. Number of omissions on the left and on the right side is recorded.